CLINICAL TRIAL: NCT06417385
Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)-Paired Breastfeeding to Improve Breastfeeding at Discharge
Brief Title: taVNS-Paired Breastfeeding to Improve Breastfeeding at Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Haley Burdge, Medical/Dental Resident, Department of Pediatrics, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00131771
Record Dates: First submitted 2024-04-19; First posted 2024-05-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Premature Birth; Breastfeeding, Exclusive; Feeding; Difficult, Newborn
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- taVNS treatment group (Experimental): All 10 infants will receive active taVNS during breastfeeding sessions. There is no randomization or blinding involved.
  Interventions: Device: taVNS soterix device

INTERVENTIONS:
Device: taVNS soterix device — Soterix is a custom modified, FDA-cleared electrical stimulator that meets the criteria of the FDA for investigational use. Neoleads will be placed in order to deliver electrical stimulation using microcurrent (<2.5mA) with breastfeeding, on with sucking and swallowing and off with rest for 5 feeds per week for 2 weeks.

SUMMARY:
Investigators aim to improve the skills of premature or sick term infants in breastfeeding by boosting motor learning with transcutaneous vagus nerve stimulation. Investigators will recruit 10 premature, ≥ 35 weeks gestational age, or convalescing sick term infants admitted to the NICU at MUSC to participate in this study. Infants will receive taVNS treatments once a day with breastfeeding's for up to 14 days. Before each treatment, the researcher will determine how much electrical stimulation is needed for the infant to feel a slight tingle without discomfort, and during daily treatment paired with breastfeeding the infant will continue to receive this level of electrical stimulation, coinciding with latching and sucking, repeated over the duration of the feed. Investigators will collect information about the pre- and post-feed weights, the length of time for each feed, and observations of latch, suck, and swallow techniques by the infant from parents and the lactation consultant. Investigators will also evaluate parental satisfaction associated with their infant's ability to breastfeed after taVNS by providing parental satisfaction surveys at the beginning, after 1 and 2 weeks, and at 3 months after the end of the study to assess infants' progress in and maintenance of breastfeeding abilities.

If the pairing of breastfeeding with taVNS is able to result in improved outcomes of effective breastfeeding in infants in the neonatal intensive care units, this intervention could be further utilized by NICUs to increase the rate of premature and sick term infants who are successfully able to breastfeed at the time of discharge and maintain breast feeding longer after discharge. This would allow premature infants to acquire the many benefits of breastmilk as well as contribute towards the strengthening of the maternal-infant bond that breastfeeding has been shown to enhance.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≥ 35 weeks post-menstrual age,
* Clinically stable, without significant respiratory support,
* Deemed safe to breastfeed by OT/SLP/lactation,
* Maternal interest in breastfeeding,
* Are not breastfeeding well despite the assistance of a lactation consultant.

Exclusion Criteria:

* Cardiomyopathy,
* Unstable bradycardia,
* Significant respiratory support,
* Absent maternal interest in breastfeeding, or infant or mother with contraindications to breastfeeding such as infantile galactosemia,
* Maternal HIV without adequate viral suppression,
* Maternal illicit drug use.

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study population will include preterm infants at ≥ 35 weeks post-menstrual age or term infants requiring NICU admission due to medical illness. The study population will also include the infants' mothers who will participate in daily breastfeeding sessions and complete parental satisfaction surveys.
Enrollment: 10 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Adequate volume transfer during breastfeeding | 2 weeks
  Measured by pre- and post-feed weights (grams)
Infant's ability to sustain breastfeeding for a length of time | 2 weeks
  Average length of active feeding at the breast (minutes)
Targeted motor learning of skills involved in breastfeeding | 2 weeks
  Demonstration of successful latch, suck, and swallow techniques by the infant per LATCH scoring (L= latch, A= audible swallowing, T= type of nipple (inverted, flat, everted after stimulation), C= Comfort of mother during feed, H= Hold/positioning of infant), scoring 0-10 (2 points per question) with 10 being the highest and optimal score.
Targeted motor learning of skills involved in breastfeeding | 2 weeks
  Demonstration of successful latch, suck, and swallow techniques by the infant by study personnel descriptions (Only lactation consultants are trained to obtain LATCH scores, thus when no lactation consultant is present, study personnel will simply describe infant's demonstrated skills during the session without a specific measurement tool)

SECONDARY OUTCOMES:
Frequency of breastfeeding assessed by study specific survey | 2 months
  Answers to related questions on taVNS-paired breastfeeding parental satisfaction survey
Parent satisfaction with infant's ability to breastfeed assessed by study specific survey | 2 months
  Answers to related questions on taVNS-paired breastfeeding parental satisfaction survey
Level of connectedness and social-emotional bond felt by mother towards infant assessed by study specific survey | 2 months
  Answers to related questions on taVNS-paired breastfeeding parental satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Haley Burdge, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Shawn Jenkins Children's Hospital, Charleston, South Carolina, United States